CLINICAL TRIAL: NCT02518464
Title: Ticagrelor Therapy for RefrACTORy Migraine Study Pilot (TRACTOR)
Brief Title: Ticagrelor Therapy for RefrACTORy Migraine Study
Acronym: TRACTOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Robert Sommer, Assistant Professor of Clinical Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAO4109
Record Dates: First submitted 2015-08-06; First posted 2015-08-07 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Migraine; Headache; Migraine Headache
Keywords: headache; chronic; migraine; right to left shunt
MeSH Terms: conditions — Migraine Disorders; Headache; Bronchiolitis Obliterans Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ticagrelor 90 mg twice per day (Experimental): Interventions include the following: All participants will have a loading dose of Ticagrelor (Brilinta) 180 mg administered in the office at the time of enrollment. Thereafter, for 28 days, Ticagrelor 90 mg tablet will be taken once in the morning and once in the evening, as close to 12 hours apart as possible. Each day, the subject will receive a text message reminder to login to the website, to record her/his headache activity.
  Interventions: Drug: Ticagrelor 90 mg twice per day

INTERVENTIONS:
Drug: Ticagrelor 90 mg twice per day — Patients will be loaded with 180 mg of Ticagrelor during the enrollment office visit and provided with a 28 day supply of Ticagrelor, 90 mg twice per day. P2Y12 reactivity unit (PRU) testing will be conducted at 7-14 days. If the patient has a positive response, they will have the option of continued access of Ticagrelor 180 mg for another 2 months. Participants will be reminded via text message daily to complete a headache survey on line in order to track their headaches.
  Other Names: Brilinta

SUMMARY:
This is a prospective, open-label, single-arm pilot study treating 40 subjects to assess the hypothesis that P2Y, G protein-coupled 12 (P2Y12) inhibition with Brilinta/ticagrelor (90 mg by mouth (PO) twice a day) reduces episodic and/or chronic migraine headache symptoms in patients with right to left shunt. Headache frequency while on Brilinta/ticagrelor will be compared with the documented baseline for each subject. If the Brilinta/ticagrelor therapy was effective (> 50% reduction in monthly headache days), the subject could elect to continue therapy for an additional two months (56 days), while continuing to complete daily headache logs.

DETAILED DESCRIPTION:
Migraine headaches are poorly understood, and can be severely debilitating. Many types of drugs have been tried in migraine sufferers including anti-depressants, anti-seizure medications, blood pressure medicines and others. The investigators have shown that in a small number of patients, a certain type of blood thinner (Clopidogrel) can reduce or eliminate migraine headaches in patients who also have a hole in the heart wall that allows flow from the right side of the heart to the left. Ticagrelor is a blood thinning drug which works in the same way as the clopidogrel, but is broken down by the body differently and thus allows everyone to use it. The investigators wish to test this medication to see if it works as well, or better than the clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* At least one year history of Episodic or Chronic migraine headache symptoms
* At least 6 headache days per month
* Subject able to complete online daily headache log

Exclusion Criteria:

* Inability to understand the study or history of non-compliance with medical advice
* Currently taking a P2Y12 inhibitor
* Known hypersensitivity to Brilinta/ticagrelor
* History of stroke/transient ischemic attack (TIA) in the previous 6 months
* Active bleeding from any site
* Active peptic ulcer disease or upper gastrointestinal (GI) bleeding within six (6) months
* Migraine onset after 50 years of age
* Renal impairment: Creatinine Clearance < 60 cc/min
* Severe hepatic impairment with total bilirubin > 3.0 mg/dL
* Thrombocytopenia with platelet count < 100,000 / ul
* History of intracranial hemorrhage
* Contraindications to blood thinner therapy or history of major bleeding episode while taking blood thinner therapy
* Need for chronic oral anti-coagulation therapy (i.e. Atrial Fibrillation)
* Need for chronic anti-platelet therapy (i.e. drug-eluting (DE) Stent), including daily aspirin use
* Need for daily nonsteroidal anti-inflammatory drug (NSAID) use
* Need for daily carbamazepine therapy or other strong CYP3A inhibitors or potent CYP3A inducers
* Need for simvastatin or lovastatin greater than 40 mg daily
* Symptomatic bradycardia or syncope
* Pregnancy or currently breast-feeding, or plan to become pregnant during the study period
* Planned surgery during the study time-frame
* Previously implanted patent foramen ovale (PFO), atrial septal defect (ASD), pacemaker, inferior vena cava filter, or left atrial appendage closure device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Sommer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reisman AM, Robbins BT, Chou DE, Yugrakh MS, Gross GJ, Privitera L, Nazif T, Sommer RJ. Ticagrelor for Refractory Migraine/Patent Foramen Ovale (TRACTOR): An open-label pilot study. Neurology. 2018 Nov 27;91(22):1010-1017. doi: 10.1212/WNL.0000000000006573. PMID 30478067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited from the hospital-based cardiology and headache clinics at Columbia University Medical Center and through the private offices of the study physicians. All subjects were evaluated by a Neurologist and fulfilled MHA criteria of the International Classification of Headache Disorders (ICHD - 3 Beta).
Period: Overall Study
Arm/Group | Ticagrelor 90 mg Twice Per Day
Started | 40
Completed | 38
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ticagrelor 90 mg Twice Per Day
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 1
  Unknown or Not Reported | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Responders
Description: A participant will be considered to have achieved the primary efficacy endpoint (a "Responder") if she/he has >50% reduction in the number of monthly headache days during the month of therapy compared with participant's own baseline. If there is < 50% reduction in the number of migraine days, she/he will be considered a Non-Responder.
Time Frame: 1 month from baseline
Measure: Count of Participants; unit: Participants
Groups:
- Ticagrelor 90 mg Twice Per Day: Interventions include the following: All participants will have a loading dose of Ticagrelor (Brilinta) 180 mg administered in the office at the time of enrollment. Thereafter, for 28 days, Ticagrelor 90 mg tablet will be taken once in the morning and once in the evening, as close to 12 hours apart as possible. Each day, the subject will receive a text message reminder to login to the website, to record her/his headache activity.
  Ticagrelor 90 mg twice per day: Patients will be loaded with 180 mg of Ticagrelor during the enrollment office visit and provided with a 28 day supply of Ticagrelor, 90 mg twice per day. P2Y12 reactivity unit (PRU) testing will be conducted at 7-14 days. If the patient has a positive response, they will have the option of continued access of Ticagrelor 180 mg for another 2 months. Participants will be reminded via text message daily to complete a headache survey on line in order to track their headaches.
  40 subjects were enrolled.
Arm/Group | Ticagrelor 90 mg Twice Per Day
Number analyzed (Participants) | 40
Participants | 17

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Ticagrelor 90 mg Twice Per Day: Two patients did not complete the TRACTOR Trial protocol due to adverse medication side effects, and five other patients had mild systemic symptoms which were potentially related to ticagrelor. Five additional patients reported unusual bruising while on ticagrelor but had no other clinical issues and completed the trial protocol. There were no significant bleeding issues in any patient treated with ticagrelor. All adverse medication effects were evaluated by the TRACTOR Trial DSMB. None were deemed to be a serious adverse event.
Arm/Group | Ticagrelor 90 mg Twice Per Day
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 10/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 90 mg Twice Per Day (N=40)
Bruising (Skin and subcutaneous tissue disorders) | 5 (5)
mild systemic symptoms (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT02518464/Prot_SAP_000.pdf